CLINICAL TRIAL: NCT06482736
Title: Effect Of Extracorporeal Shockwave Therapy on Tension-Type Headache in Adolescent Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Kerolous Ishak Shehata, lecturer, October 6 University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004547
Record Dates: First submitted 2024-06-22; First posted 2024-07-01 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Tension-Type Headache
MeSH Terms: conditions — Tension-Type Headache | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Experimental): receive exercise program for 20-30 min which include include cervical ROM to warm up,cool down, and stretching of cervical, upper thoracic spine (trapezius,levator scapula, sternocleidomastoid) and strengthening exercises (cervical isometric,concentric conctration of deep flexor muscles) each exercise consist of three sets of five to ten repetitions will be performed with 30-60S rest period between sets
  Interventions: Device: Extracorporeal Shockwave Therapy
- Study group (Experimental): receive Extracorporeal Shockwave Therapy and the same exercise program as group A, three sessions per week for 12 weeks (3 menstrual cycles).
  Interventions: Device: Extracorporeal Shockwave Therapy

INTERVENTIONS:
Device: Extracorporeal Shockwave Therapy — Extracorporeal Shockwave Therapy could reduce the pain of myofascial pain syndrome by pain signal alteration, promoting angiogenesis and increasing perfusion in ischemic tissues induced by sensitization of nociceptors and muscle ischemia.

SUMMARY:
Chronic headaches in adolescents can have consequences such as absence from school, inability to maintain social activities, and additional disorders such as anxiety, depression, problems sleeping, and reduced quality of life to investigates the efficacy shock wave diathermy on tension headaches in adolescent females

DETAILED DESCRIPTION:
The prevalence of headaches increases with age, with a prevalence of 82% during adolescence. Extracorporeal Shockwave Therapy could reduce the pain of myofascial pain syndrome by pain signal alteration, promoting angiogenesis and increasing perfusion in ischemic tissues induced by sensitization of nociceptors and muscle ischemia

ELIGIBILITY:
Inclusion Criteria:

* Suffering from chronic tension headache (headaches occur 15 or more days a month for at least three months).
* Their age will range from 15 to 18 years.
* Having a sedentary lifestyle (A weekly physical activity of < 600 MET-minutes/ week in the international physical activity questionnaire)
* Having regular menstruation (28 to 34 days).

Exclusion Criteria:

* Using oral contraceptives or
* any hormonal treatment in the previous six months.

Ages: 15 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2023-08-08 (Actual); Study Completion 2024-01-22 (Actual)

PRIMARY OUTCOMES:
digital algometer | The evaluation took place before and after 8 treatment visits using the positional inhibition technique. The treatment was carried out for 4 weeks, 2x a week, lasting 45 to 60 minutes each session.
  Measure pain intensity pre and post treatment which tested the pain points of the muscles: upper trapezius, levator scapula, sternocleidomastoid, splenius head and neck bilaterally.
Electromyography (EMG) for neck muscles | The evaluation took place before and after 8 treatment visits using the positional inhibition technique. The treatment was carried out for 4 weeks, 2x a week, lasting 45 to 60 minutes each session.
  Measure muscle activity pre and post treatmentupper trapezius, levator scapula, sternocleidomastoid, splenius head and neck bilaterally
Headache impact test questionnaire | The treatment was carried out for 4 weeks, 2x a week, lasting 45 to 60 minutes each session.
  The evaluation took place before and after 8 treatment visits using the positional inhibition technique. The treatment was carried out for 4 weeks, 2x a week, lasting 45 to 60 minutes each session.

CONTACTS AND LOCATIONS:
Overall Officials: Kerolous IS kelini, Study Director — Cairo University
Locations (1):
- Kerolous Ishak Shehata Kelini, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No